CLINICAL TRIAL: NCT06950567
Title: Evaluation of the Effectiveness of a Psychoeducational Intervention on Benzodiazepine Use in the Population Over 64 Years Old in Primary Care
Acronym: BENZOS-AP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Magi Claveria (Other)
Collaborators: Fundacio d'Atencio Primaria (Other)
Responsible Party: Sponsor-Investigator, Magi Claveria, Principal Investigator, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Organization: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4R24/159
Record Dates: First submitted 2025-04-11; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Benzodiazepines Deprescribing

STUDY DESIGN:
Intervention Model Description: The minimal intervention will consist of sending a "Benzoletter" to each participant's mailing address. This includes a personalized letter signed by their Family Doctor, an explanatory leaflet on how to gradually reduce benzodiazepine use, and infographics on sleep hygiene, stress, and anxiety.
  Among the participants, 45 will form the control group, while 24 will be part of the intervention group, which will also receive psychoeducational sessions and therapeutic exercises.
  The effectiveness of both interventions will be evaluated after six months.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (Sham Comparator): Mailing a letter by postal mail
  Interventions: Other: Control
- Experimental (Active Comparator): Mailing a letter by postal mail along with psycho-educational intervention and therapeutic activity.
  Interventions: Other: psycho-educational intervention and therapeutic activity

INTERVENTIONS:
Other: psycho-educational intervention and therapeutic activity — The objective is to provide knowledge and skills to tolerate/reduce discomfort so that they can begin to reduce or discontinue medication (BZD).
  The focus is on the effect of combined care, but the implementation of this approach is also evaluated, which will provide valuable knowledge for further health developments in Primary Care.
  Arms: Experimental
Other: Control — Sending a "Benzocarta" to each person's postal address-a personalized letter signed by their Family Doctor, an explanatory sheet on how to gradually reduce medication, and infographics on sleep hygiene, stress, or anxiety.
  Arms: control

SUMMARY:
The objective of this pragmatic, multicenter, randomized controlled clinical trial is to determine whether an educational intervention regarding benzodiazepine use can reduce the consumption and/or dosage of these drugs in individuals over 64 years old.

It aims to provide knowledge and skills to help participants tolerate or reduce discomfort, enabling them to begin decreasing or discontinuing benzodiazepine (BZD) use.

The focus is on the effect of combined care, but the implementation of this approach is also assessed, providing valuable insights for further health developments in Primary Care.

Researchers will compare a minimal intervention, consisting of sending a "Benzoletter" to each participant's mailing address, with an intensive intervention that additionally includes psychoeducational sessions and therapeutic exercises.

Participants in the intervention group will attend sessions at the Primary Care Center for a total duration of eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* People over 64 years old who have been using benzodiazepines for a period of three months or more.
* People with an active diagnosis of anxiety and/or insomnia.

Exclusion Criteria:

* People with psychiatric comorbidities, dementia, epilepsy, included in the home care program (ATDOM), institutionalized, or in palliative care.
* People with no possibility of contact or language barriers.
* People with difficulty traveling to the Primary Care Center (CAP).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 113 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants who have stopped taking benzodiazepines and/or have reduced their consumption measured in mg/week. | From the start of the intervention to six months afterward.

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Care Team of Alfarràs-Almenar., Almenar, Lleida, Spain